CLINICAL TRIAL: NCT07080489
Title: Exploring the Role of the Prefrontal Cortex in Decision-Making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: ki:elements (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-01010
Record Dates: First submitted 2025-07-10; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Depressive Disorder, Major Depressive Disorder; Healthy Volunteer; Aging
Keywords: UHF fMRI; DLPFC; fMRI; HD-tDCS; Cognitive Control; Noninvasive Brain Stimulation; Depression; Aging
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and experimentors are blinded to the intervention. The principal investigator managing randomization and code assignment is unblinded. Outcomes assessors remain blinded during data collection but will be unblinded after data collection is completed for final analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Stimulation (Healthy) (Experimental): Healthy adults aged 20 to 40 or 60 to 75 years.
  Interventions: Device: Active high-definition transcranial direct current stimulation (HD-tDCS) - anodal F3/F4
- Sham Stimulation (Healthy) (Sham Comparator): Healthy adults aged 20 to 40 or 60 to 75 years.
  Interventions: Device: Sham high-definition transcranial direct current stimulation (HD-tDCS) - anodal F3/F4
- Active Stimulation (Patient) (Experimental): Patients with mild to moderate depression aged 20 to 40 or 60 to 75 years.
  Interventions: Device: Active high-definition transcranial direct current stimulation (HD-tDCS) - anodal F3/ kathodal F4
- Sham Stimulation (Patient) (Sham Comparator): Patients with mild to moderate depression aged 20 to 40 or 60 to 75 years.
  Interventions: Device: Sham high-definition transcranial direct current stimulation (HD-tDCS) - anodal F3/ kathodal F4

INTERVENTIONS:
Device: Active high-definition transcranial direct current stimulation (HD-tDCS) - anodal F3/F4 — Participants receive anodal HD-tDCS targeting the left or right DLPFC (F3/F4).
  Arms: Active Stimulation (Healthy)
Device: Sham high-definition transcranial direct current stimulation (HD-tDCS) - anodal F3/F4 — Participants receive sham HD-tDCS targeting the left or right DLPFC (F3/F4). The device mimics the sensation of stimulation without delivering active current.
  Arms: Sham Stimulation (Healthy)
Device: Active high-definition transcranial direct current stimulation (HD-tDCS) - anodal F3/ kathodal F4 — Participants receive anodal HD-tDCS targeting the left DLPFC (F3) and cathodal stimulation targeting the right DLPFC (F4).
  Arms: Active Stimulation (Patient)
Device: Sham high-definition transcranial direct current stimulation (HD-tDCS) - anodal F3/ kathodal F4 — Participants receive sham HD-tDCS targeting the left DLPFC (F3) and right DLPFC (F4). The device mimics the sensation of stimulation without delivering active current.
  Arms: Sham Stimulation (Patient)

SUMMARY:
The goal of this study is to examine whether high-definition transcranial direct current stimulation (HD-tDCS) can influence decision-making for emotionally valenced content in younger and older adults, with or without major depression.

The main questions are:

In healthy adults, does brain stimulation modulate how people respond to emotionally valenced content during a decision-making task? What happens in the brain during modulation? Do these effects differ between younger and older adults?

In adults with depression, does brain stimulation help shift attention towards positive content during the task? What happens in the brain? Are these effects moderated by age (younger vs. older adults)?

The investigators will compare participants who receive real stimulation to those who receive sham (placebo) stimulation.

Participants will:

Receive high-definition transcranial direct current stimulation (HD-tDCS) of the dorsolateral prefrontal cortex (DLPFC)

Perform a decision-making task involving emotionally valenced words

Complete the task while undergoing a brain scan using ultra-high field 7 Tesla magnetic resonance imaging (MRI) to measure brain activity

DETAILED DESCRIPTION:
This study investigates whether non-invasive brain stimulation influences decision-making in four groups: younger adults (20-40 years) and older adults (60-75 years), healthy or with mild to moderate major depression. Participants with personality disorders or psychosis will be excluded.

The study builds on evidence that the dorsolateral prefrontal cortex (DLPFC) plays a key role in evaluating emotionally-valenced material and decision-making. The investigators will examine whether modulation of this region through high-definition transcranial direct current stimulation (HD-tDCS) affects responses to emotionally valenced information. Stimulation will be administered differently across groups based on theoretical models of hemispheric function in mood regulation.

To explore the effect of stimulation at neurotransmitter level, the investigators will use ultra-high field 7 Tesla magnetic resonance spectroscopy (MRS) to measure Gamma-aminobutyric acid (GABA) / Glutamate concentrations in regions of interest at baseline and after stimulation. This allows to examine whether changes in inhibitory/excitatory neurotransmitters are linked to altered emotional processing and decision making.

By combining brain stimulation, ultra-high field neuroimaging, and spectroscopy, this study examines how changes in brain network activity and neurotransmitter levels relate to decision-making in health and disease. The inclusion of both younger and older adults allows the investigators to explore age-related differences in these processes.

This project aims to provide mechanistic insights into decision-making in health and disease and to support the development of targeted neuromodulation therapies that could modulate emotional processing.

ELIGIBILITY:
Inclusion Criteria (Healthy):

* Written Informed Consent
* Age between 20-40 or 60-75 years
* Fluent in German
* Normal or corrected-to-normal vision
* No color blindness
* Right-handed
* Non-smoker

Exclusion Criteria (Healthy):

* History of neurological disorders
* History of psychiatric disorders
* Use of psychotropic medication
* Presence of magnetizable implants
* Alcohol or drug dependence

Inclusion Criteria (Patient):

* Written Informed Consent
* Diagnosed with mild to moderate depression
* Age between 20-40 or 60-75 years
* Fluent in German
* Normal or corrected-to-normal vision
* No color blindness

Exclusion Criteria (Patient):

* Intake of benzodiazepines or antipsychotic medication
* psychiatric disorders other than depression (e.g., psychosis, mania, personality disorders) or depression with organic cause
* Presence of magnetizable implants
* Alcohol or drug dependence

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Blood-oxygen-level-dependent (BOLD) signal changes during task-based functional magnetic resonance imaging (fMRI) | During study visit; measured continuously during the 20-minute stimulation period
  Blood-oxygen-level-dependent (BOLD) signal changes will be measured using ultra-high field functional magnetic resonance imaging (fMRI) during a cognitive decision-making task designed to engage prefrontal cortex regions associated with cognitive control and decision making. Structural T1-weighted and T2-weighted images will also be acquired for anatomical localization and normalization. Primary regions of interest (ROIs) include the dorsolateral prefrontal cortex (DLPFC), subgenual anterior cingulate cortex (sgACC), amygdala, and hippocampus.
GABA concentration (baseline) | During study visit; during a 9-minute magnetic resonance spectroscopy (MRS) session performed up to 10 minutes prior to the 20-minute stimulation period
  Magnetic resonance spectroscopy (MRS) will be used to measure Gamma-aminobutyric acid (GABA) concentrations in regions of interest at baseline. The goal is to examine stimulation-related neutransmitter changes.
GABA concentration (after stimulation) | During study visit; within 1 minute after the 20-minute stimulation period, during a 9-minute MRS scan
  Magnetic resonance spectroscopy (MRS) will be used to measure Gamma-aminobutyric acid (GABA) concentrations in regions of interest after HD-tDCS. The goal is to examine stimulation-related neutransmitter changes.
Glutamate concentration (baseline) | During study visit; during a 9-minute magnetic resonance spectroscopy (MRS) session performed up to 10 minutes prior to the 20-minute stimulation period
  Magnetic resonance spectroscopy (MRS) will be used to measure Glutamate concentrations in regions of interest at baseline. The goal is to examine stimulation-related neutransmitter changes.
Glutamate concentration (after stimulation) | During study visit; within 1 minute after the 20-minute stimulation period, during a 9-minute MRS scan
  Magnetic resonance spectroscopy (MRS) will be used to measure Glutamate concentrations in regions of interest after HD-tDCS. The goal is to examine stimulation-related neutransmitter changes.

SECONDARY OUTCOMES:
Positive Affect measured by PANAS (baseline) | During study visit; at baseline, up to two hours before the 20-minute stimulation period
  Positive Affect will be assessed using the Positive Affect subscale of the Positive and Negative Affect Schedule (PANAS). This subscale includes 10 items reflecting positive emotions. Each item is rated on a 5-point Likert scale. The sum score ranges from 10 to 50, with higher scores indicating greater levels of positive affect.
Negative Affect measured by PANAS (baseline) | During study visit; at baseline, up to two hours before the 20-minute stimulation period
  Negative Affect will be assessed using the Negative Affect subscale of the Positive and Negative Affect Schedule (PANAS). This subscale includes 10 items reflecting negative emotions. Each item is rated on a 5-point Likert scale. The sum score ranges from 10 to 50, with higher scores indicating greater levels of negative affect.
Positive Affect measured by PANAS (after stimulation) | During study visit; after stimulation, up to 1 hour
  Positive Affect will be assessed using the Positive Affect subscale of the Positive and Negative Affect Schedule (PANAS). This subscale includes 10 items reflecting positive emotions. Each item is rated on a 5-point Likert scale. The sum score ranges from 10 to 50, with higher scores indicating greater levels of positive affect.
Negative Affect measured by PANAS (after stimulation) | During study visit; after stimulation, up to 1 hour
  Negative Affect will be assessed using the Negative Affect subscale of the Positive and Negative Affect Schedule (PANAS). This subscale includes 10 items reflecting negative emotions. Each item is rated on a 5-point Likert scale. The sum score ranges from 10 to 50, with higher scores indicating greater levels of negative affect.
Storytelling (baseline) | During study visit; at baseline, up to two hours before the 20-minute stimulation period
  Participants will be asked to verbally recall one positive and one negative autobiographical memory. Verbal responses will be audio recorded and analyzed using automated speech analysis. The analysis will be performed by ki:elements, an external provider specialized in speech analysis.
Storytelling (after stimulation) | During study visit; after stimulation, up to 1 hour
  Participants will be asked to verbally recall one positive and one negative autobiographical memory. Verbal responses will be audio recorded and analyzed using automated speech analysis. The analysis will be performed by ki:elements, an external provider specialized in speech analysis.

OTHER OUTCOMES:
Verbal intelligence measured by Wortschatztest (WST) | During study visit; at baseline, up to two hours before the 20-minute stimulation period
  The Wortschatztest (WST) is a standardized test assessing verbal intelligence by measuring vocabulary knowledge in German. It is administered to account for participants' baseline language ability, helping to control for individual differences in German word knowledge that may affect performance in the decision-making task. The maximum possible score is 42, with higher scores indicating better vocabulary knowledge.
Number of (participants with) adverse effects | During study visit; after stimulation, up to 1 hour
  Participants report adverse effects using the Adverse Effects Questionnaire. They indicate the presence and severity of possible adverse effects related to transcranial direct current stimulation (tDCS), including headache, neck pain, scalp pain, tingling, itching, burning, drowsiness, and concentration difficulties. Severity is rated on a scale from none, mild, moderate, to strong. Participants also report the perceived duration of each sensation and whether they attribute it to the stimulation. Open responses for any additional sensations are collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Peter, PhD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Department of Old Age Psychiatry and Psychotherapy, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
Time Frame: Data will be shared at the end of the study on a platform of the University of Bern (Boris Portal).